CLINICAL TRIAL: NCT06241417
Title: Point-of-care Ultrasound to Evaluate Renal Prognosis of Acute Kidney Injury in Critically Ill Patients an Observational Study
Brief Title: Ultrasound to Evaluate Acute Kidney Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Associated Professor of Critical Care Medcine, Southeast University, China
Other Study IDs: 2023ZDSYLL379-P01
Record Dates: First submitted 2024-01-23; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Acute Kidney Injury; Critically Ill
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine and plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- renal recovery: Renal recovery was defined as not satisfied by AKI criteria which was defined by KDIGO.
- non renal recovery: Non renal recovery was defined by presenting at least KDIGO Stage 1 criteria or death.

SUMMARY:
Acute kidney injury is a common complication in critically ill patients. This condition can significantly prolong the length of hospital stay, increase the cost of hospitalization, and have a high mortality rate and a poor prognosis. Early assessment of patients' prognosis with acute kidney injury is vital for clinical treatment. Point-of-care ultrasound and renal injury biomarkers can be used to evaluate kidney injury at different levels. Therefore, it is speculated that dynamic monitoring can accurately predict the prognosis of patients with kidney injury.

DETAILED DESCRIPTION:
AKI is a common complication in patients with severe disease, significantly prolonging hospital stay, increasing hospital costs, high mortality, and poor prognosis. Epidemiological studies abroad have shown that the incidence of AKI in the intensive care unit (ICU) is about 39%, and the 90-day case fatality rate is 34%.

The renal prognosis of AKI is also a central concern for intensivists, as the renal prognosis also affects the long-term survival outcomes of patients with AKI. In a long-term follow-up of 1538 hospitalized patients, Bhatraju et al. found that in the AKI population, patients who did not recover their renal function during hospitalization had a significantly higher long-term mortality rate than those who recovered.

The main causes of AKI include prerenal factors, renal factors, and postrenal factors. The proportion of AKI caused by postrenal causes in ICU patients is small and can be easily treated and corrected, and prerenal and renal factors are the main causes of AKI in ICU patients. Therefore, the assessment of prerenal and nephrogenic factors in patients with AKI can predict the prognosis of AKI more accurately. An important mechanism of AKI pathogenesis is renal hypoperfusion. Urine output is often used to evaluate renal perfusion in clinical practice, but the specificity of urine output to assess renal perfusion is poor and is affected by factors such as age, stress, surgery, and diuretic use.

Point-of-care ultrasound has the advantages of non-invasive, simple, rapid, and reproducible evaluation, and has been widely used in critically ill patients. Color Doppler ultrasonography and contrast-enhanced ultrasonography can be used to measure renal perfusion parameters and assess renal function. Darmon et al. used renal ultrasound to measure the renal resistance index (RRI) and semi-quantitative renal perfusion (SQP) of renal blood flow in 371 critically ill patients and found that the RRI was significantly higher in patients with AKI than in patients without AKI, but RRI performed poorly in predicting short-term renal prognosis in AKI. Compared with two-dimensional ultrasound, contrast-enhanced ultrasound can visualize changes in renal microcirculation and provide a clearer assessment of renal perfusion. Yoon et al. performed contrast-enhanced renal sonography in 48 patients with AKI and found that the slope of renal cortex washout and peak medulla intensity predicted renal recovery, but the predictive performance was modest.

Novel biomarkers of AKI can identify kidney injury earlier, determine the severity of the injury, and assess prognosis. Komaru et al. measured urinary neutrophil gelatinase-associated lipids transport proteins (NGAL) and serum interleukin-6 levels in 133 patients with AKI requiring continuous renal replacement (CRRT) in the ICU. Urinary NGAL levels at the end of CRRT have been found to predict successful weaning of CRRT.

Based on the above research background, the following scientific hypothesis is proposed: the combination of renal ultrasound and AKI biomarkers can better predict the renal prognosis of AKI patients.

ELIGIBILITY:
Inclusion Criteria:

Meets diagnostic criteria for AKI (according to KDIGO guidelines); Age ≥ 18 years and ≤ 80 years

Exclusion Criteria:

Chronic kidney disease stage IV-V, maintenance hemodialysis; Kidney tumors; History of kidney transplantation; Nephrectomy; Pregnancy; Arrhythmias that affect the measurement of renal ultrasound.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute kidney injury patients in intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-25 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of acute kidney disease | Seven days after enrollment
  AKD was defined by presenting at least KDIGO Stage 1 criteria for >7 days after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital Affiliated to Southeast University, Nanjing, Jiangsu, China